CLINICAL TRIAL: NCT07162688
Title: Effects and Mechanism of Omega-3 Polyunsaturated Fatty Acids on Acute Graft-versus-host Disease (aGVHD) After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Effects of Omega-3 Fatty Acids on Acute Graft-versus-Host Disease After Allogeneic Stem Cell Transplantation.
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, The First Affiliated Hospital of Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Omega3-aGVHD-01; In-hospital project fund (Other Grant/Funding Number: FujianMU)
Record Dates: First submitted 2025-05-26; First posted 2025-09-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Graft-Versus-Host Disease(GVHD)
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Acute Graft-versus-Host Disease; Immunomodulation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, randomized, parallel assignment trial. Participants undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT) will be randomly assigned in a 1:1 ratio to either receive standard care or standard care plus intravenous Omega-3 lipid emulsion. The intervention will continue until hematopoietic engraftment or up to Day +35 post-transplantation. The primary objective is to assess the effect of Omega-3 supplementation on the incidence and severity of acute graft-versus-host disease (aGVHD) within 100 days post-transplant.
Masking Description: This is an open-label trial. No participants, care providers, investigators, or outcome assessors are masked to group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 Lipid Emulsion Group (Experimental): Participants in this arm will receive standard post-transplant care plus intravenous Omega-3 lipid emulsion at a dose of 2 mL/kg/day (equivalent to 0.2 g/kg of fish oil). The infusion will begin during the conditioning phase and continue daily until neutrophil and platelet engraftment or up to Day +35 post-transplantation.
  Interventions: Drug: Omega-3 Lipid Emulsion
- No Intervention (No Intervention): Participants in this arm will receive standard post-transplant care as per institutional protocol. No Omega-3 lipid emulsion or additional investigational product will be administered. This group serves as the control group for evaluating the effects of Omega-3 supplementation in the experimental arm.

INTERVENTIONS:
Drug: Omega-3 Lipid Emulsion — Intravenous Omega-3 lipid emulsion administered at a dose of 2 mL/kg/day (equivalent to 0.2 g/kg of fish oil), starting from the conditioning phase prior to hematopoietic stem cell infusion and continuing daily until neutrophil and platelet engraftment or up to Day +35 post-transplantation. The emulsion is infused over 4-6 hours and combined with medium- and long-chain triglyceride emulsion as part of parenteral nutrition.
  Other Names: ω-3 Lipid Emulsion; Omega-3 PUFA; Omega-3 Fatty Acid Emulsion
  Arms: Omega-3 Lipid Emulsion Group

SUMMARY:
Study Title:

A Study on the Effects and Mechanisms of Omega-3 Polyunsaturated Fatty Acids on Acute Graft-Versus-Host Disease (aGVHD) Following Allogeneic Hematopoietic Stem Cell Transplantation

Study Type:

Open-label, randomized, single-center proof-of-concept clinical trial

Objective:

To evaluate the immunomodulatory and metabolic effects of Omega-3 polyunsaturated fatty acids (PUFAs) in patients undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT), and to explore their potential in preventing and mitigating acute graft-versus-host disease (aGVHD).

Study Population:

More than 30 patients aged 18-65 years undergoing allo-HSCT.

Intervention:

Daily intravenous infusion of Omega-3 lipid emulsion at 2 mL/kg (equivalent to 0.2 g/kg of fish oil), administered in combination with medium/long-chain fat emulsion, starting from the conditioning regimen until neutrophil and platelet engraftment or up to Day +35.

Primary Endpoint:

Incidence and severity of aGVHD within 100 days post-transplant.

Secondary Endpoints:

Immune reconstitution (changes in T, B, and NK cell subsets) Lipid and metabolic regulation (TC, TG, HDL-C, LDL-C, TBA) Incidence and severity of infections Overall survival (OS) and progression-free survival (PFS)

Statistical Analysis:

Chi-square/Fisher's exact test, Kaplan-Meier survival analysis with log-rank test, multivariate regression, metabolomics and transcriptomics (PCA, PLS-DA), and pathway enrichment and correlation analyses.

Expected Outcome:

Omega-3 supplementation is expected to reduce the incidence and severity of aGVHD by modulating immune responses and metabolic processes, thereby providing a novel preventive strategy for post-transplant complications.

DETAILED DESCRIPTION:
This study evaluates the therapeutic potential of Omega-3 polyunsaturated fatty acids (PUFAs) in the context of acute graft-versus-host disease (aGVHD) following allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Omega-3 fatty acids have demonstrated beneficial effects on cardiovascular health, regulation of immune responses, and modulation of inflammatory pathways. Given that current immunosuppressive therapies for aGVHD are often associated with significant side effects and limited efficacy, the development of safer and more effective interventions is urgently needed.

The investigators have previously established robust research platforms, including HTLV-1 detection methods, infection and disease models (such as humanized mice and Diannan small-eared pig models), as well as multi-omics technologies covering virology, immunology, genomics, and epigenetics. Building on this foundation, the present trial aims to:

Conduct integrative analyses of viral genomic characteristics and host genetic susceptibility to construct a risk prediction model for ATL development, providing data support for clinical prevention and treatment strategies.

Characterize the dynamic spatial and temporal changes of the host immune microenvironment at the single-cell level after HTLV-1 infection, and elucidate key nodes of virus-host interaction that contribute to aGVHD pathogenesis.

Establish and optimize therapeutic strategies targeting the NPM1/B23-sHBZ interaction, and evaluate the specificity, efficacy, and safety of Omega-3 PUFA-based immunotherapy alone or in combination with agents such as PD-1 antibodies, chidamide, and DNA methyltransferase inhibitors.

Assess treatment outcomes by monitoring virological suppression, tumor burden, immune and metabolic microenvironment alterations, epigenetic modifications, incidence and severity of cytokine release syndrome (CRS), hematological parameters, and overall survival.

This proof-of-concept study is expected to provide important scientific evidence for the development of novel immunotherapy approaches targeting ATL, with the potential to improve prognosis and expand therapeutic options for patients undergoing allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT)
2. Age 18 to 65 years (inclusive)
3. Male or female
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3
5. Expected survival of at least 100 days
6. Willingness to participate and provide written informed consent

Exclusion Criteria:

1. History of solid organ transplantation
2. Serum triglycerides ≥ 7.9 mmol/L
3. Uncontrolled diabetes
4. Severe dyslipidemia (e.g., LDL-C ≥ 4.9 mmol/L)
5. Contraindications to parenteral nutrition (e.g., severe electrolyte imbalance, acidosis)
6. Severe hepatic impairment (AST/ALT > 3× ULN)
7. Creatinine clearance < 15 mL/min
8. Known allergy to Omega-3, fish, or egg protein
9. Significant psychiatric illness or substance abuse interfering with study compliance
10. Participation in another clinical trial or receipt of other experimental treatments during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Acute Graft-versus-Host Disease (aGVHD) Within 100 Days After Allogeneic Hematopoietic Stem Cell Transplantation | Within 100 days post-transplantation
  The primary outcome is to assess the incidence and clinical severity of acute graft-versus-host disease (aGVHD) occurring within 100 days following allogeneic hematopoietic stem cell transplantation. aGVHD will be diagnosed and graded based on standard clinical criteria involving skin, liver, and gastrointestinal tract involvement, using established staging and grading systems.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) at Day 100 Post-Transplantation | 100 days post-transplantation
  Progression-Free Survival (PFS) is defined as the time from transplantation to disease relapse, progression, or death from any cause, whichever occurs first. Participants who are alive and without disease progression at Day 100 will be considered progression-free.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, PhD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the exploratory nature of the study, limited sample size, and institutional data protection policies. Additionally, privacy concerns and ethical constraints prevent the public release of sensitive patient-level data.